CLINICAL TRIAL: NCT00304083
Title: Phase II Trial of Chemotherapy in Sporadic and Neurofibromatosis Type 1 Associated High Grade Malignant Peripheral Nerve Sheath Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Stage III or Stage IV Malignant Peripheral Nerve Sheath Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARC006; SARC-006; NCI-06-C-0043; NCI-P6452; UMN-2007CG077; NCT00266890 (obsolete NCT alias)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-05

CONDITIONS: Neurofibromatosis Type 1; Sarcoma
Keywords: adult neurofibrosarcoma; childhood neurofibrosarcoma; metastatic childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; stage IV adult soft tissue sarcoma; neurofibromatosis type 1
MeSH Terms: conditions — Neurofibromatosis 1; Sarcoma; Neurofibrosarcoma | interventions — Filgrastim; Doxorubicin; Etoposide; Ifosfamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy and local control by radiotherapy and surgery (Experimental): Patients receive doxorubicin hydrochloride and ifosfamide (IA) chemotherapy. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity. Patients then receive etoposide and ifosfamide (IE) chemotherapy. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also receive filgrastim (G-CSF) subcutaneously (SC) after each chemotherapy course. After recovery from chemotherapy, patients undergo radiotherapy and receive 2 more courses of IE during radiotherapy followed by 2 more courses of IA after completion of radiotherapy. Some patients may then undergo surgery.
  Interventions: Biological: filgrastim; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Procedure: conventional surgery; Radiation: radiation therapy
- Chemotherapy and local control by surgery (Experimental): Patients receive 2 courses of IA followed by 2 courses of IE as above. After recovery from chemotherapy, patients undergo surgery. After recovery from surgery, patients receive 2 more courses of IA followed by 2 more courses of IE in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: ifosfamide; Procedure: conventional surgery

INTERVENTIONS:
Biological: filgrastim — Given subcutaneously
  Arms: Chemotherapy and local control by radiotherapy and surgery
Drug: doxorubicin hydrochloride — Given IV
Drug: etoposide — Given IV
Drug: ifosfamide — Given IV
Procedure: conventional surgery — Patients undergo surgery
Radiation: radiation therapy — Patients undergo radiotherapy
  Arms: Chemotherapy and local control by radiotherapy and surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, ifosfamide, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy with or without radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating patients with stage III or stage IV malignant peripheral nerve sheath tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response rate (complete and partial) in patients with sporadic or neurofibromatosis type 1 (NF1)-associated high-grade stage III or IV malignant peripheral nerve sheath tumors (MPNSTs) after treatment with 4 courses of chemotherapy comprising doxorubicin hydrochloride and ifosfamide (IA) followed by etoposide and ifosfamide (IE).

Secondary

* Evaluate the utility of fludeoxyglucose F18 positron emission tomography (^18FDG-PET) and automated MRI volumetric tumor analysis as tools to assess response to treatment.
* Correlate response evaluation by 2-dimensional WHO criteria, 1-dimensional RECIST criteria, ^18FDG-PET, and volumetric MRI with percent necrosis in tumor specimens from patients who undergo surgery for local control after chemotherapy.
* Evaluate the response of plexiform neurofibroma(s) (if present) to chemotherapy using WHO criteria and automated volumetric MRI analysis.
* Evaluate the molecular biology of sporadic and NF1-associated MPNSTs by performing a detailed pathologic analysis of tumor samples with the goal to analyze if markers can be identified that predict for response to chemotherapy or outcome.
* Construct a tissue microarray from submitted tumor samples, that will be used in the future to identify novel targets for treatment of MPNSTs.
* Assess if a serum biomarker can be identified, that predicts for the presence of a MPNST versus benign plexiform neurofibroma.
* Increase the knowledge of the epidemiology and clinical presentation of NF1-associated MPNSTs.

OUTLINE: This is a multicenter study. Patients are stratified according to type of malignant peripheral nerve sheath tumor (MPNST) (sporadic MPNST vs neurofibromatosis type 1 [NF1]-associated MPNST). Patients receive 1 of 2 treatment regimens depending on the location of the MPNST and tumor response to chemotherapy.

* Chemotherapy and local control by radiotherapy and surgery: Patients receive doxorubicin hydrochloride and ifosfamide (IA) chemotherapy comprising doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 and ifosfamide IV over 1 hour on days 1-5. Treatment repeats every 21 days for 2 courses in the absence of unacceptable toxicity. Patients then receive etoposide and ifosfamide (IE) chemotherapy comprising etoposide IV over 1 hour and ifosfamide IV over 1 hour on days 1-5. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients also receive filgrastim (G-CSF) subcutaneously (SC) after each chemotherapy course beginning on day 6 or 7 and continuing until blood counts recover or pegfilgrastim SC once on day 6 or 7.

After recovery from chemotherapy, patients undergo radiotherapy and receive 2 more courses of IE during radiotherapy followed by 2 more courses of IA after completion of radiotherapy. Some patients may then undergo surgery.

* Chemotherapy and local control by surgery: Patients receive 2 courses of IA followed by 2 courses of IE as above. After recovery from chemotherapy, patients undergo surgery. After recovery from surgery, patients receive 2 more courses of IA followed by 2 more courses of IE in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 74 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed sporadic or neurofibromatosis type 1 (NF1)-associated high-grade malignant peripheral nerve sheath tumors (MPNSTs)

  * Stage III or stage IV (metastatic) disease
* Measurable disease, defined as at least 1 tumor that is measurable in 2 dimensions on CT scan or MRI

PATIENT CHARACTERISTICS:

* Ejection fraction normal by echocardiogram or MUGA
* Serum creatinine normal for age OR creatinine clearance > 60 mL/min
* SGPT < 5 times upper limit of normal (ULN)
* Bilirubin < 2.5 times ULN
* Absolute neutrophil count ≥ 1,500/mm^3*
* Hemoglobin ≥ 9.0 g/dL*
* Platelet count ≥ 100,000/mm^3*
* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment NOTE: * Unsupported

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for MPNST
* Prior surgical resection of MPNST allowed provided residual or recurrent measurable disease is present
* Recovered from toxic effects of all prior therapy
* At least 3 weeks since prior chemotherapy or biologic therapy for treatment of a plexiform neurofibroma, optical pathway tumor, or other NF1-associated tumor (in patients with NF1)
* At least 6 weeks since prior radiotherapy for treatment of a plexiform neurofibroma, optical pathway tumor, or other NF1-associated tumor (in patients with NF1)
* At least 4 weeks since prior radiotherapy to the area involved by MPNST
* No other concurrent growth factors (e.g., sargramostim [GM-CSF] or interleukin-11)

  * Concurrent epoetin alfa allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C. Widemann, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (17):
- United States (17):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Sarcoma Oncology Center, Santa Monica, California
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance at Washington University, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- NF1 MPNST; Sporadic MPNST: 2 cycles of ifosfamide + doxorubicin ('IA') followed by 2 cycles of ifosfamide + etoposide ('IE') prior to local control measures (surgery and/or radiation therapy).
  Local control with surgery and/or radiation will commence after recovery from toxicities. Patients, who undergo surgery only, will receive 2 more cycles of 'IA' followed by 2 cycles of 'IE' beginning after recovery from surgery. Patients, who receive radiation therapy in addition to surgery, will receive 2 cycles of 'IE' during radiation treatment, as doxorubicin cannot be concurrently administered with radiation therapy, and 2 cycles of 'IA' after completion of radiation treatment.
  1 cycle = 21 days Doxo = Doxorubicin 37.5 mg/m2/dose IV over 15 minutes on days 1, 2 Ifos = Ifosfamide 1,800 mg/m2/dose IV over 60 minutes on days 1, 2, 3, 4, 5 Etop = Etoposide 100 mg/m2/dose IV over 60 minutes on days 1, 2, 3, 4, 5
Period: Overall Study
Arm/Group | NF1 MPNST | Sporadic MPNST
Started | 34 | 14
Completed 4 Cycles | 22 | 7
Patients Treated With Surgery | 7 | 3
Patients Treated With Surgery and RT | 5 | 1
Patients Treated With RT Only | 4 | 2
Patients Had Neither RT or Surgery | 6 | 1
Completed | 12 | 6
Not Completed | 22 | 8
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 8 | 3
Not completed — Disease Progression | 5 | 1
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NF1 MPNST | Sporadic MPNST | Total
Number analyzed (Participants) | 34 | 14 | 48
Age, Continuous [Median (Full Range); unit: years] | 33 [8 to 66] | 40 [13 to 72] | 36.5 [8 to 72]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 22 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Rate (Complete Response and Partial Response)
Description: WHO criteria was used to determine responses due to the nonspherical shape of most MPNST. Complete Response (CR), Disappearance of all target lesions; Partial response (PR), >=50% decrease of target lesions.
Time Frame: After 4 Cycles (1 cycle=21 days)
Population: 37/48 patients total were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | NF1 MPNST | Sporadic MPNST
Number analyzed (Participants) | 28 | 9
Participants
  Partial response | 5 | 4
  Complete response | 0 | 0
  Stable Disease | 20 | 4
  Progressive Disease | 3 | 1

2. Secondary Outcome: Response of Plexiform Neurofibroma to Neoadjuvant Chemotherapy Using Volumetric MRI Analysis
Description: Evaluate the response of plexiformneurofibroma (if present) to neoadjuvant chemotherapy using WHO criteria and volumetric MRI analysis as a tool for response assessment
Time Frame: After 4 Cycles (1 cycle=21 days)
Population: MRI imaging of the MPNST and plexiform neurofibroma component was not sufficient to allow for volumetric analysis over time. Reasons include differences in imaging technique over time and incomplete coverage of the entire tumor.
Arm/Group | NF1 MPNST | Sporadic MPNST
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Utility of Fludeoxyglucose F18 Positron Emission Tomography (18FDG-PET) and Automated MRI Volumetric Tumor Analysis to Assess Response to Treatment
Description: Evaluate the utility of fludeoxyglucose F18 positron emission tomography (18FDG-PET) and automated MRI volumetric tumor analysis as tools to assess response to treatment.
Time Frame: After 4 cycles
Population: This assessment involved 18FDG-PET and MRI imaging of the MPNST and plexiform neurofibroma component. Due to technical issues with MRI imaging, data was not reliably collected from any study participant to allow for meaningful analysis.
Arm/Group | NF1 MPNST | Sporadic MPNST
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Response Evaluation Using WHO, RECIST, 18 FDG-PET and Volumetric MRI With Percent Necrosis in Tumor Specimens
Description: Correlate response evaluation using WHO, RECIST, 18 FDG-PET and volumetric MRI with percent necrosis in tumor specimens from patients who undergo surgery for local control after chemotherapy.
Time Frame: After 4 cycles
Population: 33 patients were evaluable for response after cycle 4, response evaluation using WHO and RECIST was performed. Response evaluation was not assessed with 18 FDG-PET and volumetric MRI.
Measure: Count of Participants; unit: Participants
Groups:
- NF1 and Sporadic MPNST: 2 cycles of ifosfamide + doxorubicin ('IA') followed by 2 cycles of ifosfamide + etoposide ('IE') prior to local control measures (surgery and/or radiation therapy).
  Local control with surgery and/or radiation will commence after recovery from toxicities. Patients, who undergo surgery only, will receive 2 more cycles of 'IA' followed by 2 cycles of 'IE' beginning after recovery from surgery. Patients, who receive radiation therapy in addition to surgery, will receive 2 cycles of 'IE' during radiation treatment, as doxorubicin cannot be concurrently administered with radiation therapy, and 2 cycles of 'IA' after completion of radiation treatment.
  1 cycle = 21 days Doxo = Doxorubicin 37.5 mg/m2/dose IV over 15 minutes on days 1, 2 Ifos = Ifosfamide 1,800 mg/m2/dose IV over 60 minutes on days 1, 2, 3, 4, 5 Etop = Etoposide 100 mg/m2/dose IV over 60 minutes on days 1, 2, 3, 4, 5
Arm/Group | NF1 and Sporadic MPNST
Number analyzed (Participants) | 33
Participants
  Responses in agreement | 29
  Responses were not in agreement | 4

5. Secondary Outcome: Perform Pathologic Analysis of Tumor Samples to Analyze the Number of Participants With Markers as Predictors of Response
Description: Evaluate the molecular biology of sporadic and NF1-associated MPNSTs by performing a detailed pathologic analysis of tumor samples with the goal to analyze if markers can be identified that predict for response to chemotherapy or outcome.
Time Frame: After 4 cycles
Population: The rows are among three different categories: Histologic Variant, Cellularity and Necrosis.
Measure: Count of Participants; unit: Participants
Arm/Group | NF1 MPNST | Sporadic MPNST
Number analyzed (Participants) | 26 | 11
Participants
  Histologic Variant- Conventional | 15 | 7
  Histologic Variant- Perineural | 1 | 0
  Histologic Variant- Epithelioid | 0 | 2
  Histologic Variant- Divergent | 1 | 0
  Histologic Variant- Mixed histology | 9 | 2
  Low Cellularity | 0 | 0
  Moderate Cellularity | 5 | 4
  High Cellularity | 21 | 7
  Necrosis- absent | 5 | 1
  Necrosis 1-10% | 8 | 2
  Necrosis 10-50% | 10 | 5
  Necrosis >50% | 3 | 3

6. Secondary Outcome: Construct Tissue Microarray to Identify Novel Targets for Treatment for the Number of Participants With Available Tissue
Description: Construct a tissue microarray from submitted tumor samples that will be used in the future to identify novel targets for treatment of MPNSTs. The tissue microarray looked at various gene deletions and amplifications.
Time Frame: After 4 cycles
Population: The number of participants vary in the rows from overall number analyzed, due to the tissue that was available for testing.
Measure: Number; unit: participants
Arm/Group | NF1 MPNST | Sporadic MPNST
Number analyzed (Participants) | 20 | 10
participants
  EGFR (7p12) amplification: number analyzed (Participants) | 20 | 8
  EGFR (7p12) amplification | 3 | 1
  TOPO2A (17q21-q22) amplification: number analyzed (Participants) | 19 | 10
  TOPO2A (17q21-q22) amplification | 5 | 2
  Her2/Neu (17q11-q12) amplification: number analyzed (Participants) | 18 | 10
  Her2/Neu (17q11-q12) amplification | 2 | 0
  Cyclin D1 (11q13) amplification: number analyzed (Participants) | 19 | 9
  Cyclin D1 (11q13) amplification | 1 | 2
  c-MYC (8q24) amplification: number analyzed (Participants) | 20 | 8
  c-MYC (8q24) amplification | 5 | 0
  N-MYC (2p24) amplification: number analyzed (Participants) | 16 | 6
  N-MYC (2p24) amplification | 3 | 1
  NF1 (17q11) deletion: number analyzed (Participants) | 19 | 9
  NF1 (17q11) deletion | 7 | 0
  p16 (9p21) deletion: number analyzed (Participants) | 14 | 6
  p16 (9p21) deletion | 10 | 3
  RB (13q14) deletion: number analyzed (Participants) | 17 | 10
  RB (13q14) deletion | 1 | 2
  p53 (17q13) deletion: number analyzed (Participants) | 19 | 9
  p53 (17q13) deletion | 6 | 2

7. Secondary Outcome: Identify the Number of Participants With a Serum Biomarker to Predict the Presence of MPNST Versus Benign Plexiform Neurofibroma
Description: Assess if a serum biomarker can be identified that predicts for the presence of a MPNST versus benign plexiform neurofibroma.
Time Frame: After 4 cycles
Population: Data looked at response evaluable patients with MPNST and focused on the TOPO2A gene being amplified.
Measure: Count of Participants; unit: Participants
Arm/Group | NF1 and Sporadic MPNST
Number analyzed (Participants) | 20
Participants
  NF1 patients with gene amplified | 3
  Sporadic patients with gene amplified | 2

8. Secondary Outcome: Provide Epidemiology and Clinical Presentation of the Number of Participants With NF1-associated MPNSTs.
Description: Increase the knowledge of the epidemiology and clinical presentation of NF1-associated MPNSTs.
Time Frame: After 4 cycles
Population: Clinical evaluation of patients with NF1 was performed at trial enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | NF1 MPNST
Number analyzed (Participants) | 34
Participants
  ≥10 subcutaneous neurofibromas | 10
  6 or more CAL: number analyzed (Participants) | 28
  6 or more CAL | 17
  Intertriginous freckling: number analyzed (Participants) | 28
  Intertriginous freckling | 19
  Neurofibromas: number analyzed (Participants) | 28
  Neurofibromas | 26
  Plexiform neurofibroma: number analyzed (Participants) | 20
  Plexiform neurofibroma | 12
  Paraspinal neurofibromas: number analyzed (Participants) | 24
  Paraspinal neurofibromas | 12
  ≥10 cutaneous neurofibromas: number analyzed (Participants) | 24
  ≥10 cutaneous neurofibromas | 13
  Optic glioma: number analyzed (Participants) | 18
  Optic glioma | 1
  Glioma: number analyzed (Participants) | 18
  Glioma | 1
  Scoliosis: number analyzed (Participants) | 22
  Scoliosis | 5
  Intellectual delay: number analyzed (Participants) | 26
  Intellectual delay | 8
  Hypertension: number analyzed (Participants) | 28
  Hypertension | 8

ADVERSE EVENTS:
Arm/Group | NF1 and Sporadic MPNST
Serious Adverse Events (participants affected / at risk) | 13/48
Other Adverse Events (participants affected / at risk) | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NF1 and Sporadic MPNST (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Anemia (Blood and lymphatic system disorders) | 4
Altered mental status (Psychiatric disorders) | 1
Aphasia (Psychiatric disorders) | 1
Somnolence (Nervous system disorders) | 4
Secondary acute myeloid leukemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NF1 and Sporadic MPNST (N=48)
Neurotoxicity (Nervous system disorders) | 3 — Eight patients had dose reductions of chemotherapy with three of those being for neurotoxicity associated with ifosfamide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No